CLINICAL TRIAL: NCT04166448
Title: LUMIERE on the PLACENTA : A Study on the Added Value of MRI
Brief Title: LUMIERE on the PLACENTA
Status: Withdrawn | Type: Observational
Why Stopped: Never start
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: LUMIERE Fondation ( fondation-lumiere.org) under the aegis of Fondation de France (Unknown); University of Paris 5 - Rene Descartes (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190335
Record Dates: First submitted 2019-09-17; First posted 2019-11-18 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: High risk IUGR patients: EPF<10th perc or PA<10th perc and Doppler ombilical IP> 95th percentile, EPF or PA<3th perc (reference curves from Collège Français d'Echographie Fœtale, between 20 et 34 GW),
  Interventions: Other: Fetal MRI
- Group 2: Low risk IUGR patients: EPF et PA>20th perc (reference curves from Collège Français d'Echographie Fœtale, between 20 et 34 GW)
  Interventions: Other: Fetal MRI

INTERVENTIONS:
Other: Fetal MRI — The MRI examination added by this research, without injection or sedation, induces no risk for the mother as for the fetus(es)

SUMMARY:
The frequency of IUGR is between 3 and 10% of births. The etiologies and mechanisms of IUGR are multiple. The placental insufficiency, that is the defect of perfusion, is, however, the principal mechanism, far in front of other maternal or fetal causes. This placental insufficiency is also now recognized as an essential risk factor for cardiovascular and metabolic diseases, such as diabetes, in adulthood. The interest in understanding in utero development is thus further increased by the short-, medium- and long-term consequences of placental dysfunction. However, there are few ways to evaluate uteroplacental vascularization in vivo. MRI is an imaging technique used routinely in the exploration of the fetus in addition to ultrasound. Its safety on the fetus and the mother is largely demonstrated at 1.5T. There are also MRI sequences used daily in the clinic to evaluate perfusion and organ structure in children and adults (brain, kidney, heart, etc.). Their application for evaluation of perfusion and placental structure, although still confined to research, is very promising. The investigator's team has extensive experience, in animals or in children, in the use of these sequences that could be used to evaluate placental function in vivo. The ASL (Arterial Spin Labeling) in particular is the most encouraging functional imaging technique because it allows today to measure an organ blood flow quantitatively and without injection of contrast medium.

DETAILED DESCRIPTION:
The inclusion will take place at the earliest at 20 weeks after the completion of the standard morphological ultrasound of the 2nd trimester (carried out at 20-24SA) and at the latest at 35 SA, within the framework of one of the 2 clinical subgroups of patients considered (high risk and low risk).

The objectives of this study will be achieved by the prospective setting up of a LUMIERE cohort on PLACENTA.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy without fetal malformation seen on ultrasound. Group 1: High risk IUGR patients

  * EPF<10th perc or PA<10th perc and Doppler ombilical IP> 95th percentile,
  * EPF or PA<3th perc reference curves from Collège Français d'Echographie Fœtale, between 20 et 34 GW,

Group 2: Low risk IUGR patients

• EPF et PA>20th perc reference curves from Collège Français d'Echographie Fœtale, between 20 et 34 GW

Exclusion Criteria:

* - Contraindication to MRI
* Impossible subsequent follow up
* Maternal status contraindicates continuation of pregnancy
* Participation in another search
* "Protected" patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant patients with low and high risk of placental IUGR followed in the Fetal Medicine Department of the Necker-Enfants Malades hospital.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Changes in placental blood flow as seen in vascular IUGR | From inclusion to end of neonatal period (max 25 weeks)
  25% reduction in overall placental perfusion measured ASL with IUGR (defined as <3th perc birth weight) versus controls (birth weight> 10th perc)

SECONDARY OUTCOMES:
Placental response to maternal oxygenation (BOLD) | From inclusion to end of neonatal period (max 25 weeks)
  BOLD effect
structural changes of the placenta | From inclusion to end of neonatal period (max 25 weeks)
  Diffusion coefficient (ADC)
structural changes of the placenta | From inclusion to end of neonatal period (max 25 weeks)
  T2 * mapping
Measurement of placental volume | From inclusion to end of neonatal period (max 25 weeks)
  Placental segmentation
Measurement of IUGR by fetal segmentation (MRI), | From inclusion to end of neonatal period (max 25 weeks)
  Fetal volume
evaluation of brain resonance | From inclusion to end of neonatal period (max 25 weeks)
  BOLD effect, - ADC coefficient and IVIM parameters by variation of T2 * relaxation time
evaluation of kidney resonance | From inclusion to end of neonatal period (max 25 weeks)
  BOLD effect, - ADC coefficient and IVIM parameters by variation of T2 * relaxation time
evaluation of liver resonance | From inclusion to end of neonatal period (max 25 weeks)
  BOLD effect, - ADC coefficient and IVIM parameters by variation of T2 * relaxation time
Reproducibility of the examination analysis | After study completion, an average of one year
  Correlations between microcirculatory parameters in utero, fetal weight at MRI and birth weight
Uterine arteries | From inclusion to end of neonatal period (max 25 weeks)
  Measurement of blood flow in the uterine arteries by MRI 4D FLOW (in development) and Doppler (US) (feasibility study)
Acceptability of the examination for the patient: questionnaire | at IRM examination
  Will be assessed by a questionnaire given to pregnant women after the MRI,
Acceptability of the examination for the patient: Likert scale | at IRM examination
  will be assessed once by a Likert scale: 4 points Likert (poor, average, good, very good)
Specific Absorption Rate for each type of sequence | From inclusion to end of neonatal period (max 25 weeks)
  SAR measurement (Specific Absorption Rate)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Salomon, MD, PhD, Principal Investigator — Principal Investigator
Locations (1):
- Necker - Enfants Malades Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No